CLINICAL TRIAL: NCT06753708
Title: Evaluation of the Nutritional Status of Patients Hospitalized in the Palliative Care Unit and Receiving Tube Enteral Nutrition Support
Brief Title: Evaluation of the Nutritional Status of Palliative Care Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Zehra Margot Celik, Principal Investigator, Marmara University
Other Study IDs: 16.09.2024/85
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-12

CONDITIONS: Palliative Care; Tube Feeding
Keywords: Palliative Care; Malnutrition; Nutritional Status; Tube Feeding
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Palliative Care Patients: Patients over 18 years of age who received inpatient treatment in the Palliative Care Clinic of a State Hospital

SUMMARY:
This study evaluates the nutritional status of palliative care patients receiving enteral tube feeding. It aims to assess their condition using nutritional screening tools, anthropometric measurements and biochemical data to improve standards of care, patient safety and outcomes. The study will take place at a state hospital palliative care clinic from November 2024 to March 2025, with a possible extension to June 2025.

Participants will be adults aged 18 years and older undergoing enteral tube feeding. Informed consent will be obtained, and data collection will include in-person interviews, patient questionnaires, food consumption records completed by family members, and biochemical data from medical records. Nutritional information will be analyzed using BeBIS software, and SPSS will be used for statistical analysis.

The study aims to create effective nutrition plans, improve clinical protocols, and improve healthcare outcomes. By addressing gaps in the literature, particularly regarding enteral tube feeding in palliative care, this research will benefit patients, families, healthcare providers, and institutions. Anticipated benefits include improved patient care, reduced complications, shorter hospital stays, and cost savings to the healthcare system.

DETAILED DESCRIPTION:
The data obtained from food consumption records will be transferred to the Nutrition Information System (BeBIS) program by the researcher and total energy, macro and micronutrients will be calculated. The data of the individuals participating in the study will be analyzed with SPSS 28.0 (Statistical Package for Social Sciences for Windows) statistical package program.

Institutional, social and economic benefits are also among our goals with this research. The institutional benefits of the research include the evaluation of the nutritional status of patients receiving tube enteral nutrition support, the creation of effective nutrition plans and, when necessary, the provision of improvement recommendations.In addition, by reviewing and updating clinical enteral nutrition protocols, standards of care will be improved and patient safety will increase. This process will encourage more efficient use of resources and increase knowledge and awareness of enteral nutrition among healthcare professionals. It will contribute to the organization's quality improvement efforts, support performance assessments in nutrition and patient care, and improve patient satisfaction and treatment outcomes through effective nutrition support. The societal benefits are to contribute to improving national and international standards for patients receiving tube enteral nutrition support through the development of more effective and targeted nutrition strategies in patient care, efficient use of resources, education on nutrition management for health professionals, families and caregivers, and the development of nutrition management policies based on research findings. The economic benefits of the research will be achieved by improving the nutritional status of patients, reducing complication rates and shortening hospital stays with the effective implementation of tube enteral nutrition management. This will result in a significant reduction in healthcare costs and encourage more efficient use of resources. As a result, reduced material and labor costs will contribute to a more sustainable model of care by reducing the financial burden on the healthcare system.This research aims to evaluate the nutritional status of patients hospitalized in a palliative care ward and receiving tube enteral nutrition support using anthropometric measurements, nutrition screening tools, scales and biochemical findings. Although there are similar studies in the literature, there is no study that specifically examines the status of tube enteral nutrition in palliative care. Existing studies generally focus on enteral nutrition support, deficiencies or malnutrition and quality of life in palliative care. Considering the increase in the elderly population and the number of palliative care hospitalizations, this study aims to make an important contribution to the existing gap in the literature.

The study is planned to include patients over 18 years of age who received inpatient treatment in the Palliative Care Clinic of a Hospital between November 2024 and March 2025 and who received tube enteral nutrition. Approval was obtained from Marmara University Institute of Health Sciences Non-Interventional Clinical Research Ethics Committee for the conduct of this study. A power analysis was performed with the Epi-Info program and the sample size was determined as 132 participants. Considering the losses, 145 patients will be included in the study. If the targeted sample size is not reached, the data collection process is planned to be extended until June 2025. Verbal and written informed consent will be obtained from the patients before data collection. All patients who agree to participate in the study will be interviewed face-to-face and the questionnaire form will be filled out by the researcher. The questionnaire form will include sections on general information about the patient, medical nutrition therapy, anthropometric measurements and biochemical parameters. In addition, each patient's relatives will be asked to fill in the food consumption record form. The nutrition screening tools NRS-2002 and GLIM Criteria will be applied to each patient by the investigator. Filling out the enteral nutrition record form and taking anthropometric measurements will be done by the investigator. Biochemical findings required for the study will be obtained from patient files.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being treated in the Palliative Care Clinic
* Being fed with one of the tube enteral nutrition methods (only enteral/enteral + oral/enteral)

Exclusion Criteria:

* Having any limb amputation
* Being hospitalized in the Palliative Care Clinic for less than 3 days
* Receiving parenteral nutrition support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Palliative Care patients from a State Hospital in Istanbul / Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Malnutrition Status - NRS-2002 Score | 7 days after admission to the palliative care unit
  The NRS-2002 tool will be used to evaluate the malnutrition risk of patients. This screening tool, developed by ESPEN in 2002, includes components for nutritional status and disease severity. The total score will be recorded based on the assessment conducted by the researcher.
  Unit of Measure: NRS-2002 score; >3 indicates malnutrition.
Body Mass Index (BMI) | 7 days after admission to the palliative care unit
  Calculated from weight (measured or estimated) and height (measured or estimated).
  Unit of Measure: kg/m²
Upper Mid-Arm Circumference | 7 days after admission to the palliative care unit
  Measured using a flexible tape measure. Unit of Measure: cm
Skinfold Thickness | 7 days after admission to the palliative care unit
  Measured at specified anatomical sites using a Saehan Medical Skinfold Caliper. Unit of Measure: Millimeters (mm)]
Enteral Nutrition Record | 7 days after admission to the palliative care unit
  For each patient, enteral nutrition method, type, total daily feeding hours and nutrition infusion rate will be recorded on the form. Interruptions in enteral nutrition due to medical, technical or patient-related reasons, duration of interruption and treatment changes will also be recorded. This information will be obtained from the patients' nutrition files after obtaining the necessary permissions. Target energy and protein levels will be calculated by the investigator for each patient.
Food Consumption Record | 7 days after admission to the palliative care unit
  A 24-hour food consumption record will be obtained for patients with oral intake in addition to tube enteral nutrition.
Nutritional Biomarker Index | 7 days after admission to the palliative care unit
  A composite nutritional biomarker index will be calculated based on laboratory findings that have been recorded in patients files in the last 7 days. The index will include hemoglobin, hematocrit, albumin, and prealbumin levels, combined using a weighted scoring system to reflect overall nutritional status.
  Unit of Measure: Composite score (unitless)

SECONDARY OUTCOMES:
Phenotypic Criteria - Weight Loss | 7 days after admission to the palliative care unit
  Percentage of weight loss will be calculated and recorded. Unit of Measure: Percentage (%)
Phenotypic Criteria - Body Mass Index (BMI) | 7 days after admission to the palliative care unit
  BMI will be determined using weight and height measurements. If direct measurements are not feasible due to patient bedridden status, height will be estimated from knee length, and weight will be calculated using upper mid-arm circumference and calf circumference measurements through validated equations.
  Unit of Measure: BMI (kg/m²)
Phenotypic Criteria - Muscle Mass | 7 days after admission to the palliative care unit
  Muscle mass will be estimated using a specific validated method (e.g., bioelectrical impedance analysis or anthropometric measurements).
  Unit of Measure: Muscle mass (kg)
Etiologic Criteria - Food Intake | 7 days after admission to the palliative care unit
  Daily food intake will be assessed based on a standardized dietary questionnaire or other method. Unit: Kilocalories per day (kcal/day)
Etiologic Criteria - Inflammatory Status | 7 days after admission to the palliative care unit
  Inflammatory markers (e.g., CRP, albumin) will be measured using laboratory analysis.
  CRP levels (mg/L), albumin (g/dL)
Knee Length | 7 days after admission to the palliative care unit
  Knee length will be measured using a specialized caliper for bedridden patients.
  Unit of Measure: Centimeters (cm)
Calf Circumference | 7 days after admission to the palliative care unit
  Calf circumference will be measured using a flexible measuring tape. Unit of Measure: Centimeters (cm)
Height | 7 days after admission to the palliative care unit
  Height will be directly measured if feasible, or estimated from knee length using validated equations for bedridden patients.
  Unit of Measure: Meters (m)
Body Weight | 7 days after admission to the palliative care unit
  Body weight will be measured directly if feasible, or estimated using upper mid-arm circumference and calf circumference measurements through validated equations.
  Kilograms (kg)
Hemoglobin | 7 days after admission to the palliative care unit
  Hemoglobin levels will be recorded from patient files. Unit of Measure: g/dL
Hematocrit | 7 days after admission to the palliative care unit
  Hematocrit levels will be recorded from patient files. Unit of Measure: Percentage (%)
Platelet Count | 7 days after admission to the palliative care unit
  Platelet Count will be recorded from patient files. Unit of Measure: ×10³/μL
Leukocyte Count | 7 days after admission to the palliative care unit
  Leukocyte Count will be recorded from patient files. Unit of Measure: ×10³/μL
Neutrophil Count | 7 days after admission to the palliative care unit
  Neutrophil Count will be recorded from patient files. Unit of Measure: ×10³/μL
Lymphocyte Count | 7 days after admission to the palliative care unit
  Lymphocyte Count will be recorded from patient files. Unit of Measure: ×10³/μL
Blood Urea Nitrogen (BUN) | 7 days after admission to the palliative care unit
  BUN levels will be recorded from patient files. Unit of Measure: mg/dL
Creatinine | 7 days after admission to the palliative care unit
  Creatinine levels will be recorded from patient files. Unit of Measure: mg/dL
Magnesium | 7 days after admission to the palliative care unit
  Magnesium levels will be recorded from patient files. Unit of Measure: mg/dL
Sodium | 7 days after admission to the palliative care unit
  Sodium levels will be recorded from patient files. Unit of Measure: mmol/L
Potassium | 7 days after admission to the palliative care unit
  Potassium levels will be recorded from patient files. Unit of Measure: mmol/L
Chlorine | 7 days after admission to the palliative care unit
  Chlorine levels will be recorded from patient files. Unit of Measure: mmol/L
Calcium | 7 days after admission to the palliative care unit
  Calcium levels will be recorded from patient files. Unit of Measure: mg/dL
CRP | 7 days after admission to the palliative care unit
  CRP levels will be recorded from patient files. Unit of Measure: mg/L
Albumin | 7 days after admission to the palliative care unit
  Albumin levels will be recorded from patient files. Unit of Measure: g/L
Prealbumin | 7 days after admission to the palliative care unit
  Prealbumin levels will be recorded from patient files. Unit of Measure: mg/dL
Glomerular Filtration Rate (GFR) | 7 days after admission to the palliative care unit
  GFR levels will be recorded from patient files. Unit of Measure: mL/min/1.73m²

CONTACTS AND LOCATIONS:
Overall Officials: Zehra M Celik, Study Director — Marmara University
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University, Faculty of Health Sciences, Istanbul, Maltepe
  - Marmara University, Istanbul, Maltepe

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.